CLINICAL TRIAL: NCT03933072
Title: Evaluation of the Possibility of Induction of Functional Axon Regeneration in Patients With Complete Spinal Cord Injuries Using Autologous Bulbar Olfactory Ensheathing Cells and Techniques of Bridging of the Spinal Cord.
Brief Title: Autologous Bulbar Olfactory Ensheathing Cells and Nerve Grafts for Treatment of Patients With Spinal Cord Transection
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nicholls Spinal Injury Foundation (Other)
Collaborators: Wroclaw Medical University (Other); Akson, Neuro-Rehabilitation Center for the Treatment of Spinal Cord Injuries (Unknown); University College, London (Other); Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Pawel Tabakow, Ass. Professor, MD PhD, Wroclaw Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Wroclaw Walk Again Project
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Spinal Cord Injury at C5-Th10 Level With Complete Lesion; Spinal Cord Transection
Keywords: complete spinal cord injury, spinal cord transection, olfactory ensheathing cells, olfactory fibroblasts, Glial Neuropatch, nerve grafts
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: interventional study, parallel assessment, open label, non-randomized, safety-efficacy study; sponsored clinical trial;
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with complete spinal cord injury (Experimental): the planned interventions have been described in the section below
  Interventions: Procedure: obtaining of autologous human olfactory bulb, autologous sural nerve preparation; Biological: production of Glial Neuropatch; Procedure: microsurgical reconstruction of the transected spinal cord with autologous Glial Neuropatch-nerve bridges

INTERVENTIONS:
Procedure: obtaining of autologous human olfactory bulb, autologous sural nerve preparation — The operative procedure will be aimed to obtain one of the patient's olfactory bulbs. The operation will be performed using a minimally invasive intracranial microsurgical endoscopy-assisted or transnasal endoscopic approach. During the same operation the patient sural nerve will be prepared for a future grafting.
Biological: production of Glial Neuropatch — The human autologous olfactory ensheathing glia and olfactory fibroblast isolated from the olfactory bulb will be used for production of Glial Neuropatch in a laboratory facility in accordance with good manufacture procedures (GMP). The final Product will consist of the aforementioned cell suspension embedded with collagen scaffold. The European Medicines Agency/Committee for Advanced Therapies (EMA/CAT) considers that the Product Glial Neuropatch falls within the definition of a tissue engineered product of an advanced therapy medicinal product (decision EMA/CAT/293903/2018 from 22 June 2018: Scientific recommendation on classification of advanced therapy medicinal products Article 17 - Regulation (EC) No 1394/2007).
Procedure: microsurgical reconstruction of the transected spinal cord with autologous Glial Neuropatch-nerve bridges — The surgery will consists of laminectomy/laminotomy, midline durotomy above the area of spinal cord lesion, detethering of the spinal cord from fibrotic adhesions, resection of the posttraumatic spinal cord glial scar, delivering of cultured OEC/ONFs explants (Glial Neuropatch) to the area of spinal cord injury and finally bridging of the spinal cord gap by harvested autologous sural nerve grafts.

SUMMARY:
The purpose of this experimental therapy is to evaluate the safety and efficacy of transplantation of autologous olfactory ensheathing cells (OECs) and olfactory nerve fibroblasts (ONFs) obtained from the olfactory bulb with simultaneous reconstruction of the posttraumatic spinal cord gap with peripheral nerve grafts, in patients with chronic complete spinal cord injury. The treatment will be performed in two patients that have sustained an anatomically complete spinal cord transection between the spinal cord segments C5 and Th10.

All patients wanting to participate in this study have to send their application at the address:

walk-again-project.org

DETAILED DESCRIPTION:
The "Wrocław Walk Again" project is a continuation of the innovative experimental therapy involving reconstruction of patient's severed spinal cords, using their own olfactory glial cells from the olfactory bulb as well as implants from peripheral nerves. The first operation of its kind was performed in 2012. The reconstruction of the cord was a success: the patient regained partial feeling and volitional mobility in paralysed limbs (Cell Transplantation, Vol. 23, pp. 1631-1655, 2014). The experiment's success provided inspiration to continue with the project in order to assess the safety and effectiveness of the therapy applied. The continuation involves planning to qualify two patients with traumatic spinal cord injury, who will then be given treatment and physiotherapy. The programme will be conducted in Wroclaw, Poland, by an interdisciplinary team of doctors and scientists. The Nicholls Spinal Injury Foundation (UK) will be making a significant contribution to the project. Due to this, participants will not need to pay for their experimental treatment or physiotherapy.

The main goal of the study is to answer the question if there is possible to evoke functional regeneration of severed spinal cord axons after a two-stage surgical intervention in patients sustaining a complete spinal cord transection between the spinal cord segments C5 and Th10. Patients with clinically, electrophysiologically and radiologically features of complete spinal cord injury will undergo an 8-month neurorehabilitation regimen. Patients who will not show electrophysiological and clinical signs of recovery from the spinal cord injury will enter the surgical part of the study.

During the first surgery the patient's own olfactory bulb will be obtained. The human autologous olfactory ensheathing glia and olfactory fibroblast isolated from the olfactory bulb will be used for production of Glial Neuropatch in accordance with the methodology adjusted in grant number GR-797/NCN/2013 and 2012/06/M/NZ4/00138, in a laboratory facility, in accordance with the good manufacture procedures (GMP). The final Product will consist of the aforementioned cell suspension embedded with collagen scaffold. The European Medicines Agency/Committee for Advanced Therapies (EMA/CAT) considers that the Product Glial Neuropatch falls within the definition of a tissue engineered product of an advanced therapy medicinal product (decision EMA/CAT/293903/2018 from 22 June 2018: Scientific recommendation on classification of advanced therapy medicinal products Article 17 - Regulation (EC) No 1394/2007).

The second surgery will consist of laminectomy/laminotomy, midline durotomy above the area of spinal cord lesion, detethering of the spinal cord from fibrous adhesions, resection of the posttraumatic spinal cord glial scar, delivering of cultured OEC/ONFs explants (Glial Neuropatch) to the area of spinal cord injury and finally bridging of the spinal cord gap by harvested autologous sural nerve grafts.

After discharge from the hospital, the patients will be subjected to a minimum 2-year neurorehabilitation in accordance with the same program as before the operation.

ELIGIBILITY:
Inclusion Criteria:

1. A single spinal cord injury between vertebral levels C5-Th10 with a total anatomic disruption of continuity.
2. Myelopathy not exceeding 2 spinal cord segments as confirmed by MRI.
3. Complete loss of sensory and motor function below the injury, confirmed in serial control clinical studies (ASIA Category A) and neurophysiological studies (MEP, SSR, EPT, EMG, ENG, von Frey's filaments)
4. Age from 16 to 65 years.
5. Patient undergoing continuous rehabilitation.
6. Good patient motivation and cooperation, no mental disturbances.
7. Patient is ready to stay with an accompanying person for at least 3 years in Poland.
8. Patient without cardiac disease and without epilepsy, does not have peacemaker or any electronic or ferromagnetic implants.

Exclusion Criteria:

1. A coexisting lesion of the nervous system.
2. Progressive post-traumatic syringomyelia.
3. Significant spinal stenosis or instability.
4. Muscle atrophy or joint ossifications.
5. Severe systemic disease such as neoplasm, contagious disease, diabetes etc.
6. Chronic sinusitis destroying the paranasal sinuses, tumors of nasal cavities or patients with hyposmia in repetitive smell perception tests will be excluded.
7. Implants or the health status described in point 8 (see above).

Note: All patients wanting to participate in this study have to send their application via the walk-again-project.org recruitment website!

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
improvement of the neurologic state measured by the American Spinal Injury Association (ASIA) score. | up to 2 years postoperatively
  A positive outcome will be defined as any detectable improvement of motor and /or sensory function below the level of spinal cord injury, that will result that the patient will change from being with complete spinal cord injury (assigned as ASIA A) to incomplete (ASIA B,C,D or E). ASIA E means complete recovery from spinal cord injury-no clinical evidence of neurological impairment.
improvement of the strenght of trunk muscles measured by the Berg Balance scale | up to 2 years postoperatively
  a set of tests evaluating the risk of patient to fall during sitting, standing and transfers
  The results from the specific tests assign the patients to the following three groups:
  41-56 points = low fall risk; 21-40 pts. = medium fall risk, 0 -20 pts. = high fall risk
  An improvement of the trunk muscle strenght that will transfer the patient from the high fall risk group to the medium or low fall risk group will be considered as essential clinical improvement.
improvement of neurologic state measured with tests of deep sensation | up to 2 years postoperatively
  deep pressure tests applied to the specific dermatomal areas,0 points means no deep sensation while 1 point means sensation of same feeling when pressure is applied
improvement of neurologic state measured with tests of vibration | up to 2 years postoperatively
  vibration tests applied on the shoulder, elbow, wrist,finger,knee,malleolus and toe
  0 Zero, A Diminished, B More vague description - less accurate than A, C Causalgia, 2 Normal
improvement of neurologic state measured with tests of joint position sense | up to 2 years postoperatively
  joint position test applied on the wrist, thumb, little finger, knee, ankle and great toe
  0 points- absence of joint position sense (during 8 of 10 or more attempts)
  1. point- impaired sense (correct only on large movements of the joint during 8 of 10 attempts, and incorrect on small movements of the joint (8 of 10 or more attempts)
  2. points- normal sense (during 8 of 10 or more attempts) on small and large movements;

SECONDARY OUTCOMES:
decrease of muscle spasticity for at least 1 level measured the Ashworth scale | tested monthly for at least 2 years postoperatively
  The 5 level spasticity Ashworth scale includes:
  level 0- no increase in muscle tone, level 1- slight increase in muscle tone, manifested by a catch and release or by minimal, resistance at the end of the range of movement (ROM) when the affected part(s) is moved in flexion or extension, level 2-slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the reminder (less than half) of the ROM, level 3-more marked increase in muscle tone throughout most of the ROM but affected part(s) easily moved, level 4-considerable increase in muscle tone passive, movement difficult, level 5-affected part(s) rigid in flexion or extension
Spinal Cord Assessment Tool for Spastic Reflexes ( SCATS) | tested monthly for at least 2 years postoperatively
  a test evaluating the clonus rate, and the rate of flexors and extensor muscle spasms
  Clonus is rated on a 4 point scale that ranges from:
  0 No reaction
  1. Mild lasting <3sec
  2. Moderate lasting 3-10 seconds
  3. Severe lasting > 10 seconds
  Flexor spasms are rated on a 4 point scale that ranges from:
  0 No reaction
  1. Mild, less than 10 degrees of excursion in flexion at knee and hip, or extension of the great toe
  2. Moderate = 10-30 degrees of flexion at knee and hip
  3. Severe with >30 degrees of hip and knee flexion
  SCATS extensor spasms assessment 0 No reaction
  1. Mild lasting <3sec
  2. Moderate lasting 3-10 seconds
  3. Severe lasting > 10 seconds
  Test interpretation: The better the patient improvement is, the lower points he will be assigned, reaching at the end the ideal state of being without clonus and muscle spasms (0 points).
improvement of locomotion ability in the Walking Index for Spinal Cord Injury (WISCI II) test, | tested monthly for at least 2 years postoperatively
  The WISCI II test assesses the patient walking ability from being unable to walk (0 level) to being able to walk normally without any help (level 20).
  Interpretation of the test: Any patient improvement that will assign him to a higher level of walking independency compared to the preoperative state will be considered as positive outcome.
10 meter walking test | tested monthly for at least 2 years postoperatively
  a test measuring the velocity of walking the distance of 10 meters; (only the middle 6 meters are timed);
  Any improvement of the ambulation velocity will be considered as positive outcome.
2 minutes walking test | tested monthly for at least 2 years postoperatively
  a test measuring the distance ambulated in 2 minutes [m]
  Any improvement of the distance of ambulation in the period of 2 minutes will be considered as positive outcome.
time up and go test | tested monthly for at least 2 years postoperatively
  The patient should sit on a standard arm chair, placing his/her back against the chair and resting his/her arms chair's arms. Any assistive device used for walking should be nearby. Regular footwear and customary walking aids should be used. The patient should walk to a line that is 3 meters (9.8 feet) away, turn around at the line, walk back to the chair, and sit down.
  Any decrease of the time needed for completion of this test will be considered as positive outcome.
improvement measured by the spinal cord independence measure (SCIM III) test | tested monthly for at least 2 years postoperatively
  improvement of the patient self care ability
neurophysiological evidence of reconnection of fibers from motor origin | tested every 3 months for at least 2 years postoperatively
  a set of tests evaluating the conductivity of efferent central and peripheral nerve fibers and the muscle response to electrical stimulation, including motor evoked potentials (MEP), electromyography (EMG) and electroneurography (ENG),
neurophysiological evidence of reconnection of fibers from sensory origin | tested every 3 months for at least 2 years postoperatively
  the electrical perceptual thresholding (EPT) test- evaluating the dermatomal sensation of the upper and lower limbs in the condition of low voltage current application (from 0 to 7-8 mA)
  Interpretation of the test: any tingling sensation reported by the patient in the previously anesthetic dermatomes, in the condition of current below 4 mA will be considered as essential improvement of skin sensation.
neurophysiological evidence of reconnection of fibers from vegetative origin | tested every 3 months for at least 2 years postoperatively
  skin sympathetic response (SSR)
  Electrophysiological study assessing the integrity of the supraspinal autonomic pathways. Is performed on the median and tibial nerves.
  Test interpretation: any positive vegetative response in the tested paralyzed limbs that was previously absent will be considered as positive outcome.
improvement of urination registered in the urodynamic study | tested every 3 months for at least 2 years postoperatively
  a test measuring the electrophysiological activity of the bladder muscles and the bladder sensation
  Test interpretation: Any evidence of bladder detrusor -urethral sphincter synergy, together with the evidence of improved urination will be considered as positive outcome
evidence regrowth of spinal cord fibers detected on MRI scans, evidence of functional reorganization of the brain detected in advanced MRI protocols; lack of tumorigenesis, spinal cord inflammation, progressive syringomyelia; | MRI imaging of the spinal cord and brain will be performed every 3 months in the first year and every 6 months in the second year
  evidence of spinal cord fiber reconstitution and brain center reorganization detected on MRI scans, including advanced imaging techniques

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Tabakow, MD PhD, Principal Investigator — Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

REFERENCES:
- [Background] Tabakow P, Raisman G, Fortuna W, Czyz M, Huber J, Li D, Szewczyk P, Okurowski S, Miedzybrodzki R, Czapiga B, Salomon B, Halon A, Li Y, Lipiec J, Kulczyk A, Jarmundowicz W. Functional regeneration of supraspinal connections in a patient with transected spinal cord following transplantation of bulbar olfactory ensheathing cells with peripheral nerve bridging. Cell Transplant. 2014;23(12):1631-55. doi: 10.3727/096368914X685131. Epub 2014 Oct 21. PMID 25338642
- [Background] Tabakow P, Jarmundowicz W, Czapiga B, Fortuna W, Miedzybrodzki R, Czyz M, Huber J, Szarek D, Okurowski S, Szewczyk P, Gorski A, Raisman G. Transplantation of autologous olfactory ensheathing cells in complete human spinal cord injury. Cell Transplant. 2013;22(9):1591-612. doi: 10.3727/096368912X663532. PMID 24007776
- [Background] Collins A, Li D, Liadi M, Tabakow P, Fortuna W, Raisman G, Li Y. Partial Recovery of Proprioception in Rats with Dorsal Root Injury after Human Olfactory Bulb Cell Transplantation. J Neurotrauma. 2018 Jun 15;35(12):1367-1378. doi: 10.1089/neu.2017.5273. Epub 2018 Mar 29. PMID 29285976
- [Background] Ibrahim A, Li D, Collins A, Tabakow P, Raisman G, Li Y. Comparison of olfactory bulbar and mucosal cultures in a rat rhizotomy model. Cell Transplant. 2014;23(11):1465-70. doi: 10.3727/096368913X676213. Epub 2013 Dec 30. PMID 24380436
- [Background] Czyz M, Tabakow P, Hernandez-Sanchez I, Jarmundowicz W, Raisman G. Obtaining the olfactory bulb as a source of olfactory ensheathing cells with the use of minimally invasive neuroendoscopy-assisted supraorbital keyhole approach--cadaveric feasibility study. Br J Neurosurg. 2015 Jun;29(3):362-70. doi: 10.3109/02688697.2015.1006170. Epub 2015 Feb 7. PMID 25659961
- [Background] Czyz M, Tabakow P, Gheek D, Mis M, Jarmundowicz W, Raisman G. The supraorbital keyhole approach via an eyebrow incision applied to obtain the olfactory bulb as a source of olfactory ensheathing cells--radiological feasibility study. Br J Neurosurg. 2014 Apr;28(2):234-40. doi: 10.3109/02688697.2013.817534. Epub 2013 Jul 19. PMID 23869574